CLINICAL TRIAL: NCT06989775
Title: EnCompass Clamp and the AtriClip in Box Lesion and Left Atrial Appendage EXclusion Procedure for the Prevention of New Onset of Atrial Fibrillation
Brief Title: BoxX-NoAF Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CP-2024-02
Record Dates: First submitted 2025-05-12; First posted 2025-05-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-05

CONDITIONS: Post Operative Atrial Fibrillation; Atrial Fibrillation, Postoperative
Keywords: Post operative AF; Clinical AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment (Experimental): Index cardiac surgery + Ablation + Left Atrial Appendage Exclusion with AtriClip
  Interventions: Device: Isolator® Synergy™ EnCompass® Ablation System and AtriClip® LAA Exclusion System
- Control (No Intervention): Index cardiac surgery only

INTERVENTIONS:
Device: Isolator® Synergy™ EnCompass® Ablation System and AtriClip® LAA Exclusion System — Box lesion ablation with the Isolator Synergy EnCompass Clamp System and LAAE using the AtriClip LAA Exclusion System at the time of planned cardiac surgery
  Arms: Treatment

SUMMARY:
Post Operative Atrial Fibrillation (POAF) is the most common complication of cardiac surgery. POAF incidence can exceed 50% depending on the patient baseline characteristics and surgery type. Patients with POAF tend to have worse acute and long-term clinical outcomes. BoxX-NoAF is a randomized trial to evaluate if prophylactic ablation and exclusion of the Left Atrial Appendage at the time of other routine cardiac surgery can reduce the incidence of post operative AF and clinical AF during long term follow up in patients who have not yet developed AF but are at risk.

ELIGIBILITY:
Inclusion Criteria:

* Planned and clinically indicated for cardiac surgical procedure requiring cardiac bypass and opening of the pericardium
* Age ≥ 65 years and CHA2DS2-VASc ≥ 3

Exclusion Criteria:

* Documented history of atrial fibrillation or atrial flutter anytime prior to the cardiac surgery
* Prior procedure involving opening the pericardium or entering the pericardial space
* Patients undergoing off-pump surgery
* Prior LAA occlusion, exclusion, or removal (surgical or percutaneous)
* Presence of a permanent pacemaker
* Infiltrative cardiomyopathies (i.e. amyloidosis)
* Planned cardiac surgical procedure using non-sternotomy approaches
* Patients whose planned procedure is a heart transplant or implantation of any long-term ventricular assist devices
* Presence of ventricular arrhythmia
* Active endocarditis
* NYHA Class IV heart failure symptoms
* Preoperative need for an intra-aortic ballon pump or intravenous inotropes
* Active systemic infection at the time of cardiac surgery requiring antibiotics
* Known allergy to Nitinol or nickel sensitivity
* Known medical condition with expected survival of less than 1 year
* Other comorbidities that in the Investigator's opinion make the subject unsuitable candidate to complete the protocol required intervention or visits
* Current enrollment in an investigation or trial or an investigational devices or investigational drug that would interfere with this trial
* Mental impairment or other psychiatric conditions which may not allow the patient to understand the nature, significance, and scope of the trial.
* Pregnancy
* Known severe symptomatic carotid disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 30 days post index cardiac surgical procedure
  The occurrence of clinically relevant post operative AF (POAF)
Primary Safety Endpoint | 30 days post index cardiac surgical procedure
  The composite of the following events:
  * All cause Mortality
  * Reoperation
  * Deep sternal wound infection
  * Permanent stroke
  * Prolonged ventilation
  * Renal failure
  * 30-day readmission
  * Atypical left atrial flutter
  * Phrenic nerve palsy
  * Major Bleeding

SECONDARY OUTCOMES:
Powered Secondary Effectiveness Endpoint | 3 years post index cardiac surgical procedure
  The time to first occurrence of clinical atrial fibrillation from 30 days after index cardiac surgical procedure through 3-years

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Morton Plant Hospital - BayCare Health System, Inc., Clearwater, Florida
  - St. Joseph's Hospital - BayCare Health System, Inc., Clearwater, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Wellstar Health System, Marietta, Georgia
  - Corewell Health, Grand Rapids, Michigan
  - Ascension Saint Thomas, Nashville, Tennessee
- Hamilton General Hospital, Hamilton, Ontario, Canada